CLINICAL TRIAL: NCT01716832
Title: Effectiveness of Mindfulness Walking on Stress Reduction
Brief Title: Walking for Stress Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Benno Brinkhaus, Prof. MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Walking_Stress_Reduction
Record Dates: First submitted 2012-10-24; First posted 2012-10-30 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Healthy Subjects

ARMS (2):
- Mindfulness walking (Experimental)
  Interventions: Behavioral: Mindfulness Walking
- No intervention (waiting list) (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness Walking — Mindful walking in a small group twice a week for 60 minutes within 4 weeks.
  Arms: Mindfulness walking

SUMMARY:
The effectiveness of a mindfulness walking program is tested in subjects with a high level of subjectively perceived stress.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between 18 and 65 years
* Increased level of stress (visual analog scale >40 mm (0-100))

Exclusion Criteria:

* Regular walking training in the last 6 weeks
* Medical therapy with psychopharmacological drugs
* Regular mindfulness based meditations/exercises in the last 6 weeks
* CAM therapies against stress in the last 6 weeks
* medium or severe chronic diseases
* Stress due to chronic diseases
* Acute disease at inclusion
* Not being able to walk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Cohens Perceived Stress Scale 14 Items | 4 weeks

SECONDARY OUTCOMES:
Quality of Life (SF 36) | Baseline, 4 weeks, 12 weeks
Subjective Stress Level (Visual Analogue Scale) | Baseline, 4 weeks, 12 weeks
Assessment of effect on a Likert - Scale | 4 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Berlin, Berlin, Germany